CLINICAL TRIAL: NCT03346889
Title: Vertigo Symptoms, Balance and Vestibular Function in Patients With Vestibular Schwannoma
Brief Title: Vestibular Outcomes in Vestibular Schwannoma
Acronym: VOVS
Status: Active, not recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/765 C
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Vestibular Schwannoma
Keywords: vestibular evoked myogenic potentials; head impulse testing; quality of life
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have shown that vertigo is the symptoms that mostly affect quality of life in patients with vestibular schwannoma. There is still limited knowledge as to why some patients with this disorder develop vertigo, while others with the same diagnosis do not. The purpose of this study is to measure symptom-related quality of life and to relate this to objective disease characteristics at baseline.

DETAILED DESCRIPTION:
This is a longitudinal observational study with data collected at baseline and after treatment.

Variables collected at baseline include age, sex, tumor size, location, type (cystic/solid), tumor side, symptom variables including Dizziness Handicap Inventory, Vertigo Symptom Scale Short Form, Haukeland Dizziness Questionnaire, Visual analog scale, Hospital Anxiety and Depression Scale, RAND-12, dynamic posturography, video-based head impulse test, bithermal caloric tests, ocular and cervical vestibular evoked myogenic potentials.

Follow-up data after 1 year are the same patient-reported outcomes as at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients living i Norway referred to Haukeland University Hospital due to newly diagnosed, untreated vestibular schwannoma

Exclusion Criteria:

* Inability to undergo test protocol due to physical or language barriers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in Norway with newly diagnosed vestibular schwannoma (VS) are referred to Haukeland University Hospital for evaluation. The size of the study population therefore depends on the incidence of VS in Norway and the inclusion period. The incidence of VS in Norway is approximately 150 per year in a population of 5.2 million.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-04-23 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | Baseline and 1-year follow-up
  25-item symptom score 0 - 100 points on dizziness handicap severity

SECONDARY OUTCOMES:
Vertigo Symptom Scale Short Form | Baseline and 1-year follow-up
  15-item symptom score 0 - 60 points on vertigo symptom quality
Haukeland Dizziness Questionnaire (HDQ-10) | Baseline and 1-year follow-up
  10-item symptom score 0 - 30 points on vertigo symptom severity
Vertigo Visual Analog Scale | Baseline and 1-year follow-up
  100 mm visual analog scale on vertigo symptom severity
Hospital Anxiety and Depression Scale (HADS) | Baseline and 1-year follow-up
  14-item anxiety and depression score 0 - 42 points
RAND-12 | Baseline and 1-year follow-up
  12-item health-related quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Frederik K Goplen, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No